CLINICAL TRIAL: NCT03747835
Title: Meal-Based Exposure and Response Prevention in Anorexia Nervosa: Reducing Physiological and Self-reported Food-Related Anxiety
Brief Title: Meal-Based Exposure and Response Prevention in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Hilda and Preston Davis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00174855
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure and Response Prevention (Active Comparator): Inpatients will be provided three 90-minute sessions of Exposure and Response Prevention therapy each week.
  Interventions: Behavioral: Exposure and Response Prevention
- Motivational Interviewing (Active Comparator): Inpatients will be provided two 60-minute sessions of Motivational Interviewing each week.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Exposure and Response Prevention — Exposure and Response Prevention involves collaboratively developing a list of food-related fears with the patient and planning treatment sessions in which the patient is exposed to the fear and inhibits safety behaviors. The explicit goal of these exposure sessions will be to violate the patient's expectation regarding the feared stimulus, rather than to reduce fear.
  Arms: Exposure and Response Prevention
Behavioral: Motivational Interviewing — Motivational interviewing techniques including reflective listening to demonstrate empathy and understanding, asking questions to elicit change talk (speech that is "pro-change"), evaluating the decisional balance, and managing or "rolling with" resistance will be incorporated throughout the treatment sessions.
  Arms: Motivational Interviewing

SUMMARY:
Patients with anorexia nervosa (AN), a serious psychiatric disorder, exhibit restricted dietary intake and endorse fear of consuming calorie-dense foods, which in turn drives weight loss. Premorbid anxious personality traits and comorbid anxiety disorders are common in patients with AN. Although intensive behavioral treatment programs can achieve weight restoration in a majority of adults with AN, relapse rates are high. Predictors of relapse include elevated state anxiety and low dietary variety, including lower intake of fat, after discharge, which suggests that relapse following weight restoration may be related to inadequate fear extinction to high energy density (ED) foods during treatment and consequent resumption of restrictive eating patterns. Despite evidence of anxiety's role in the onset and maintenance of restricted eating behavior, utilizing exposure and response prevention (EX-RP) and meal-based interventions to reduce food-related fears is understudied. EX-RP is the gold standard of treatment for Obsessive Compulsive Disorder (OCD). This proposal aims to test the efficacy of an adjunct meal-based EX-RP intervention to reduce food-related fears during intensive behavioral weight restoration in hospitalized patients with AN in comparison to a control treatment, Motivational Interviewing. The investigators will assess changes in a) self-reported anxiety regarding consumption of high-ED foods, b) physiological (skin conductance and heart rate variability) responses to imagined consumption of food items elicited utilizing a visual food cue task, and c) caloric intake of a challenging test meal pre- and post-treatment. A secondary aim is to assess the relationship of early treatment response to EX-RP, operationalized as a reduction in self-reported anxiety within the first three weeks of treatment, and end-of-treatment as well as six-month post-discharge outcomes. Helping patients tolerate food-related anxiety and increase dietary variety across meal contexts may augment treatment effectiveness in adult patients during intensive treatment for AN and has potential to decrease relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM) -5 criteria for AN or Other Specified Feeding and Eating Disorder.
* Body Mass Index (BMI) > 14.0 kg/m2 and < 20.0 kg/m2
* Age > 12 years, < 66 years
* Fluency in the English language

Exclusion criteria:

* Diagnosis of schizophrenia, schizophreniform disorder, bipolar illness (type I) with active psychotic symptoms
* History of traumatic brain injury with current impairment in functioning
* Current use of benzodiazepines, as these medications may alter psychophysiological assessment
* Allergy to dairy products or chocolate contained in the test meal

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Physiological Anxiety in Response to Food Images as assessed by Skin Conductance Response | Pre-treatment and post-treatment up to 10 weeks
  Participants will view images of low- and high-ED foods, and of office products for 8 seconds each. Skin Conductance Response (microsiemens) will be recorded from electrodes placed on the palmar surface of the middle phalanges of the 2nd and 3rd fingers on the non-dominant hand.
Change in Physiological Anxiety in Response to Food Images as assessed by Heart rate variability | Pre-treatment and post-treatment up to 10 weeks
  Participants will view images of low- and high-ED foods, and of office products for 8 seconds each. Heart rate variability will be measured using ECG electrodes placed in a diagonal axis across the heart region, with a reference electrode on the stomach.
Change in amount of high calorie diet consumption | At week 2 of treatment and at discharge, up to 10 weeks
  Patients will be asked to consume a meal (1,066 kcal) consisting of calorie dense foods over a period of 45 minutes. Total caloric intake will be measured by weighing food items prior to and following the meal and identifying the proportion of the meal in kcal consumed.

SECONDARY OUTCOMES:
Change in food related anxiety as assessed by the Food Anxiety Questionnaire. | Weekly up to 10 weeks
  Patients will complete the Food Anxiety Questionnaire, which asks patients to rate their anxiety regarding consumption of 35 frequently consumed foods, using Subjective Units of Distress. Subjective Units of Distress range from 0-100, with '0' indicating no distress or anxiety and '100' indicating the highest possible level of distress or anxiety.
Change in food Choice Preferences as assessed by The Food Choice Task | Pre-treatment and post-treatment up to 10 weeks
  The Food Choice Task is a computer based task that assesses preference for low- versus high-fat food items. Patients rate food items on tastiness and healthiness and are then asked to make a series of choices regarding food preferences. The proportion of high-fat food choices made is an indication of the patient's preference for low-versus high-fat foods. A higher proportion of trials on which individuals select the high-fat food is associated with an increased willingness to consume those foods.
Eating Disorder Examination Questionnaire Scores | Pre-treatment and post-treatment up to 10 weeks
  Patients will complete the 28-item Eating Disorder Examination Questionnaire, which includes four subscales: Eating Concern, Weight Concern, Restraint, and Shape Concern. Scores on these subscales range from 0 to 7, with higher scores indicative of more pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen C Schreyer, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No